CLINICAL TRIAL: NCT05747976
Title: Genetic Disorders of Obesity Program Database
Acronym: GDOP
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie Sisley, Associate Professor, Baylor College of Medicine
Other Study IDs: H-44596
Record Dates: First submitted 2022-11-11; First posted 2023-02-28 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Childhood; Genetic Disease
MeSH Terms: conditions — Pediatric Obesity; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study collects data on children with severe, early-onset obesity.

DETAILED DESCRIPTION:
Children and adolescents who have suffered from severe weight gain prior to 5 years of age and who are seen in the Genetic Disorders of Obesity Program at Texas Children are asked to participate in a prospective, observational study. The investigators collect demographic information, body measurements, medical/family history, as well as other questionnaires. Additionally, genetic information, medical lab results, and responses to treatment options are collected. The goal of the study is to determine if the investigators can better understand which children would benefit from testing and further workup as well as to understand how obesity develops in these children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* For individuals 2 years and older, BMI > 97 percentile
* For individuals < 2 years old, weight-to-length ratio > 95th percentile

Exclusion Criteria:

* No other exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with early-onset, severe obesity.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of genetic causes of severe, early-onset obesity | through study completion, an average of 10 years
  We will measure the number of genetic variants identified in clinical testing

SECONDARY OUTCOMES:
Change in BMI over time | through participant completion, an average of 2 years
  BMI in kg/m2 will be documented over time. BMI is calculated using weight and height

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No